CLINICAL TRIAL: NCT06787950
Title: A Phase I/IIa Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Anti-tumor Activity of ASN-3186 in Patients with Advanced Solid Tumors.
Brief Title: Clinical Study of ASN-3186 in Patients with Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Yahong Meditech Co., Ltd aka Asieris (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YHGT-ASN-3186-ST-101
Record Dates: First submitted 2024-12-05; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Escalation (Experimental): Participants will receive ASN-3186 in sequential cohorts of increasing doses.
  Interventions: Drug: ASN-3186
- Dose Expansion (Experimental): Recommended doses from dose escalation stage will be studied to determine RP2D.
  Interventions: Drug: ASN-3186
- Tumor-specific Cohort Expansion (Experimental): RP2D will be further studied in tumor-specific cohorts.
  Interventions: Drug: ASN-3186

INTERVENTIONS:
Drug: ASN-3186 — ASN-3186 will be administered orally.
  Arms: Tumor-specific Cohort Expansion
Drug: ASN-3186 — ASN-3186 will be administered orally.
  Arms: Dose Escalation
Drug: ASN-3186 — ASN-3186 will be administered orally.
  Arms: Dose Expansion

SUMMARY:
This is a Phase I/IIa, open-label, multi-center, dose-escalation, and expansion study to evaluate the safety, tolerability, PK and preliminary anti-tumor activity of ASN-3186 when given orally in subjects with advanced solid tumors

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or females aged ≥ 18 years at time of signing informed consent form (ICF). Signed ICF must be obtained before the performance of any protocol-specified procedures.
2. Life expectancy ≥12 weeks evaluated by investigator.
3. ECOG Performance Score 0 to 2.
4. Histologically or cytologically confirmed advanced solid tumors defined as unresectable locally advanced or metastatic and do not have standard treatment available, or have disease progression on/after standard treatment, or cannot tolerate standard treatment.
5. For Phase Ia subjects: Subjects who have confirmed deleterious or suspected deleterious germline or somatic BRCAm, or HRRm, or HRD positive or other alterations are preferred, but gene alteration state is not mandatory as an inclusion criterion and no need to wait for biomarker detection results before enrollment.
6. For Phase Ib subjects: Subjects must have confirmed deleterious or suspected deleterious germline or somatic BRCAm, or HRRm, or HRD positive or other alterations.
7. For Phase IIa subjects: Subjects must have confirmed deleterious or suspected deleterious germline or somatic BRCAm, or HRRm, or HRD positive or other alterations.

Key Exclusion Criteria:

1． Treatment with any of the following:

1. . Prior treatment with any USP1 inhibitors.
2. . Prior treatment with radiotherapy, chemotherapy, targeted therapy or endocrine therapy within 4 weeks prior to the first dose of ASN-3186.
3. . Participated and received investigational therapy or used an investigational device or participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks or 5 × t1/2, whichever is longer, prior to the first dose of ASN-3186.

2．Subjects who expect to require any other form of anti-tumor therapy during the treatment period. 3． Subjects who have unresolved toxicity greater than common terminology CTCAE V5.0 Grade 1 from prior anti-tumor therapy prior to the first dose of ASN-3186, except for alopecia and chemotherapy-induced peripheral neurotoxicity ≤ CTCAE V5.0 Grade 2. 4． Subjects who have undergone surgery on vital organs (other than aspiration biopsy) or suffered major trauma within 4 weeks prior to the first dose, or subjects who have not recovered from any surgical effect at screening, or subjects who are scheduled for major surgery during the study period. 5． Subjects who have gastrointestinal disorders that will affect oral administration or affect the absorption of ASN-3186 as judged by the investigator. Or subjects who have severe or clinically significant gastrointestinal disease (e.g., refractory diarrhea, intractable vomiting, colitis, etc.) within 4 weeks prior to the first dose of ASN-3186 and did not recover to CTCAE V5.0 Grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2029-03-20 (Estimated); Study Completion 2029-09-20 (Estimated)

PRIMARY OUTCOMES:
phase 1( Dose Escalation Stage): Dose Limiting Toxicity (DLT) | During the first 26 Days
  DLT will be defined as toxicities that meet pre-defined severity criteria(according to the NCI CTCAE v5.0 toxicity assessment criteria),
phase 1( Dose Escalation Stage): Recommended phase 2 dose(RP2D) | 14 months
  RP2D is recommended based on MTD, safety data , efficacy data, and clinical pharmacokinetic (PK) characteristics
phase 2a: ORR | 26 months
  ORR assessed by investigators.

SECONDARY OUTCOMES:
phase1:PK characteristics | 14 months
  Plasma PK characteristics and metabolite PK characteristics of ASN-3186 after single or multiple oral administration
phase1: QT/QTc | 14 months
  To evaluate the effect of ASN-3186 on QT/QTc interval in patients with advanced solid tumors
phase1: ECG | 14 months
  To evaluate other electrocardiogram(ECG) parameters of ASN-3186 in patients with advanced solid tumors
phase1+2a：AE | 28 days after the last administration
  The occurrence of all adverse events (AE).
phase1+2a：Serious adverse events (SAE) | 28 days after the last administration
  The occurrence of all serious adverse events (SAE)
phase1+2a: Disease Control Rate（DCR） | 14months
  Disease Control Rate defined as the rate of CR+PR+SD
phase1+2a： DOR | 14 months
  duration of response(DoR）：The time during study treatment from the first tumor assessment of CR or PR to the first assessment of disease progression or all-cause death
phase1+2a: CBR | 14 months
  clinical benefit rate (CBR): Proportion of patients whose best response was observed to be CR, PR, or SD (duration ≥24 weeks) over the study period
phase1+2a: PFS | 14 months
  progression-free survival(PFS): From the date of first study treatment to the time of disease progression or all-cause death
phase1+2a: OS | 14 months
  overall survival(OS):From the date of first study treatment to the time of all-cause death
phase1+2a: biomarker | 14 months
  Relationship between biomarker and efficacy

IPD SHARING:
Plan to Share IPD: No